CLINICAL TRIAL: NCT04431674
Title: Novel Magnetic Resonance Imaging -Guided Ultrasound-Stimulated Microbubble Radiation Treatment for Patients With Chest-Wall and Locally Advanced Breast Cancer
Brief Title: Novel MRI-Guided Ultrasound Stimulated Microbubble Radiation Treatment for Patients With Chest-wall and Breast Cancer
Acronym: USmBRT-B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Senior Scientist, MD, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 077-2019
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Focused ultrasound; Microbubbles
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Prospective, Single-Centre, Single-Arm, Non-Randomized, Phase-I MRI-Guided Ultrasound Stimulated Microbubbles Radiation Treatment for Patients with Chest Wall and Breast Cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MRg-FUS MB Treatment (Experimental): Patients with locally advanced breast cancer (LABC) and chest wall tumours will receive MRI-guided ultrasound-stimulated microbubble-treatment combined with radiotherapy on a LINAC.
  Interventions: Drug: Definity Suspension for Injection

INTERVENTIONS:
Drug: Definity Suspension for Injection — MRI-guided ultrasound-stimulated microbubble-treatment

SUMMARY:
The objective of this study is to demonstrate the feasibility of novel MRI-guided ultrasound stimulated microbubble treatment to enhance radiation effects in humans receiving external beam radiotherapy delivered using a LINAC (linear accelerator) radiation therapy device.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate the feasibility of novel MRI-guided ultrasound stimulated microbubble treatment to enhance radiation effects in humans receiving external beam radiotherapy delivered using a LINAC (linear accelerator) radiation therapy device. The investigators have previously demonstrated that ultrasound and microbubble mediated endothelial cell perturbation can significantly enhance the effectiveness of radiation. It enhances tumour response to radiation significantly by synergistically destroying tumour blood vessels. The technique is targeted spatially and achieves tumour specificity by confining the low-power ultrasonic fields that stimulate microbubbles to the tumour location only. By perturbing the tumour vasculature and activating specific genetic pathways, the technique sensitizes the targeted tissues to the subsequent therapeutic application of radiation, resulting in significantly enhanced cell killing. The primary aim of this research is to evaluate the safety profile of MRI-guided ultrasound stimulated microbubble treatment and radiation in patients with chest wall and breast cancer. The secondary aim is to evaluate tumor (primary and/or nodal) response to MRg-FU + MB and radiation, as measured radiologically within the treated therapeutic regions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* All biopsy-confirmed invasive ductal, invasive lobular and other rare histologic types of carcinoma
* Patients with early stage Breast cancer, or LABC ; i.e., Stage IIA - IIIC cancers (T2 N0 M0 to Any T, N3, M0) or Stage IV (Any T, Any N, M1) per AJCC guidelines (8th Edition)
* Assessed by a multidisciplinary team of treating medical, surgical and radiation oncologist and found suitable for the treatment
* Patient referred for palliative radiotherapy or standard radiotherapy, which may include any of the following dose regimens: 1) 20 Gy in 5 fractions, 2) 30 Gy in 10 fractions, 3) 40 Gy in 10 fractions, 4) 50 Gy in 20 fractions, 5) 60 Gy in 30 fractions and 6) 66 Gy in 33 fractions.
* Able to understand and give informed consent
* Weight < 140 kg
* Target lesion accessible for MRg-FU+MB procedure
* Able to communicate sensation during the procedure
* Creatinine within normal institutional limits or creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional upper limit of normal.

Exclusion Criteria:

* Pregnant or lactating women may not participate due to the embryotoxic effects of protocol treatment. Women/ men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Unable to have a contrast-enhanced MRI scan - standard of care criteria
* Patients on anthracycline or taxane based chemotherapy
* Patients with metallic or breast implants
* Subjects with inflammatory breast cancer, connective tissue disorder, musculoskeletal deformity
* Target lesion causing ulceration, bleeding or discharge of the overlying skin
* A fibrotic scar along the proposed FU beam path
* Severe cardiovascular, neurological, renal or hematological chronic disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≥ 3
* Any condition in the investigator's opinion precludes participation
* Bleeding disorders/ High risk for deep vein thrombosis
* Unable to tolerate required stationary position during treatment
* Allergic to Definity microbubbles
* Cardiac disease or unstable hemodynamics including myocardial infarction within six months, unstable angina, congestive heart failure, ejection fraction < 50%, cardiac shunts, cardiac arrythmia and cardiac pacemaker.
* Contraindication to perflutren including subjects with a family or personal history of QT prolongation or taking concomitant medications known to cause QTc prolongation like cisapride, erythromycin, tricyclic antidepressants, Class IA and III antiarrhythmic agents and some antipsychotics like haloperidol, droperidol, quetiapine, thioridazine, ziprasidone.
* QT prolongation observed on screening ECG (QTc > 450ms for men or >470ms for women)
* Severe hypertension (diastolic BP > 100 mmHg)
* History of bleeding disorder, coagulopathy
* Severely impaired renal function with estimated glomerular filtration rate < 30ml/min/1.73m2 and/or on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity and adverse events using MRg-FUS+MB treatment in patients with chest-wall and locally advanced breast cancer | 90 days
  Incidence of toxicity and adverse events

SECONDARY OUTCOMES:
Radiological Response | 90 days
  The secondary endpoint is radiological response in breast cancer following MRg-FU + MB + radiation, after a 3 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gregory Czarnota, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moore-Palhares D, Dasgupta A, Saifuddin M, Anzola Pena ML, Prasla S, Ho L, Lu L, Kung J, McNabb E, Sannachi L, Vesprini D, Chen H, Karam I, Soliman H, Szumacher E, Chow E, Gandhi S, Trudeau M, Curpen B, Stanisz GJ, Kolios M, Czarnota GJ. Radiation enhancement using focussed ultrasound-stimulated microbubbles for breast cancer: A Phase 1 clinical trial. PLoS Med. 2024 May 17;21(5):e1004408. doi: 10.1371/journal.pmed.1004408. eCollection 2024 May. PMID 38758967
- [Derived] Dasgupta A, Saifuddin M, McNabb E, Ho L, Lu L, Vesprini D, Karam I, Soliman H, Chow E, Gandhi S, Trudeau M, Tran W, Curpen B, Stanisz G, Sahgal A, Kolios M, Czarnota GJ. Novel MRI-guided focussed ultrasound stimulated microbubble radiation enhancement treatment for breast cancer. Sci Rep. 2023 Aug 21;13(1):13566. doi: 10.1038/s41598-023-40551-5. PMID 37604988